CLINICAL TRIAL: NCT01697475
Title: An Motivational Text Messaging Walking Program for Older African Americans
Brief Title: Text-Messaging to Motivate Walking in Older African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AJPM 12-0206-126R
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Last update posted 2012-10-02 (Estimated); Status verified 2011-09

CONDITIONS: Physical Activity; Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Motivational text messaging
  Interventions: Behavioral: Motivational text messaging
- Control Group (No Intervention): Step count

INTERVENTIONS:
Behavioral: Motivational text messaging — Motivational text messaging was given for participants in the intervention group - 3 times a day, 3 times a week, for 6 weeks
  Arms: Intervention Group

SUMMARY:
This study examined the impact of using a motivational mobile text messaging intervention to increase step count among older community-dwelling African Americans. Secondary aims were to study the effects of text messaging on self-reported leisure time exercise behavior.

Hypothesis:

Participants in the motivational mobile text messaging group will have an increase step count after 6-weeks.

DETAILED DESCRIPTION:
Background: Older minority populations can benefit from increased physical activity, especially walking. Text messaging interventions have the potential to encourage positive changes in health behavior in these groups.

Purpose: To examine if a six week program of motivational text messaging increases physical activity (step count) among older African Americans in an urban setting.

Design: Randomized, controlled trial pilot study with assignment to motivational text messaging group or a control group.

Setting/Participants: Thirty-six African Americans aged 60 to 85.

Intervention: The intervention group received motivational text messages three times a day, three days a week, for six weeks. Both groups received pedometers and walking manuals to record step counts. Study was conducted and analyzed in 2011.

Main Outcome Measures: Primary outcome measure was step count. Secondary outcome measure was perceived activity levels assessed by the Leisure Time Exercise Questionnaire (LTEQ).

Results/Conclusion: In press - American Journal of Preventive Medicine (Jan 2013)

ELIGIBILITY:
Inclusion Criteria:

* African American community-dwelling adults aged 60 to 85 who were recruited from senior centers.
* had to be healthy (no restrictions and medical clearance to walk)
* had to have a mobile phone with text messaging capability

Exclusion Criteria:

* (a) any physical, psychological illness, or medical problems that restricted them from walking; (b) did not own a mobile phone with text messaging capability; or (c) were not willing or able to follow study procedures.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure was step count | 6-weeks
  Motivational text messaging led to greater improvements in step count (+679 vs. +398; P < .05)

SECONDARY OUTCOMES:
Secondary outcome measure was perceived activity levels assessed by the Leisure Time Exercise Questionnaire (LTEQ). | 6-weeks
  Motivational text messaging led to greater improvements perceived activity levels (P < .05) than the group who did not receive any text messages.

CONTACTS AND LOCATIONS:
Overall Officials: Bang Kim, PhD, Principal Investigator — Georgetown University; Karen Glanz, PhD, Study Director — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Kim BH, Glanz K. Text messaging to motivate walking in older African Americans: a randomized controlled trial. Am J Prev Med. 2013 Jan;44(1):71-5. doi: 10.1016/j.amepre.2012.09.050. PMID 23253653